CLINICAL TRIAL: NCT06910618
Title: A Multicenter Prospective Observational Study on Vertebral Fracture Risk Stratification in Patients With Vertebral Metastases
Acronym: Valid-METASTRA
Status: Not yet recruiting | Type: Observational
Sponsor: Buda Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: EUMET-101080135
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Vertebral Metastases; Vertebral Fracture
Keywords: vertebral metastasis; cancer; fracture; risk stratification
MeSH Terms: conditions — Spinal Fractures; Neoplasms; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with vertebral metastasis in ThL region: Patient diagnosed with a metastatic tumor in the thoracic and/or lumbar spine (one or more vertebral metastases in the spinal region between T1 and L5 vertebrae)

SUMMARY:
Vertebral fracture is a common clinically significant skeletal related event in cancer patients. Stratification of patients diagnosed with one or more vertebral metastases according to the risk of pathological fracture is an unresolved problem despite the fact that fractures strongly influence the quality of life (QoL) and also the overall survival. The multidimensional nature and the strong patient specificity of the risk for fracture have not been considered in previously published risk estimation models and these methods were developed and validated only on retrospective data focusing on prevalence of life-time fracture which is not really relevant at the time of the diagnosis of a vertebral metastasis. To overcome these shortcomings, the METASTRA models (METASTRA-AI and METASTRA-VPH) and the decision support system (METASTRA-DSS) are developed considering the highest possible level of patient specificity to stratify the individuals according to their risk for fracture in a clinically considerable period (within next 6 months). The prospective data collection and analysis will provide reliability and validity results on the performance of METASTRA tools as well as structured information on user's experience helping the future integration of the developed patient-specific stratification tool into the everyday clinical practice.

The study is a prospective clinical data collection from minimum 200 patients to determine the validity (i.e. Precision) in fracture risk stratification of the METASTRA-AI and METASTRA-VPH computational models and to determine the reliability of METASTRA-AI and METASTRA-VPH as well as human decision making process in patient stratification.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older
* Patient diagnosed with a metastatic tumor in the thoracic and/or lumbar spine (one or more vertebral metastases in the spinal region between T1 and L5 vertebrae)
* Min. 1 vertebra is potentially unstable based on SINS score (SINS is 7-12) and it has not been surgically stabilized previously (level of interest - LOI)
* Adjacent vertebrae are not surgically stabilized at the time of the enrollment
* Patient willing to complete 6-month follow-up
* Patient is willing and able to provide written informed consent after the nature of the study has been explained:

  * Ability to understand the content of the patient information/ ICF
  * Willingness and ability to participate in the study according to the protocol
  * Signed and dated EC approved written informed consent

Exclusion Criteria:

* Poor general status at baseline (Karnofsky scale less than 40%)
* Expected life expectancy is less than 3 months at baseline
* Spinal infection
* Ongoing litigation
* Participation in investigational clinical study at the same time or within 3 months
* Vertebral lesion/metastasis from a hematologic condition (e.g. multiple myeloma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with a metastatic tumor in the thoracic and/or lumbar spine (one or more vertebral metastases in the spinal region between T1 and L5 vertebrae)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
new vertebral fracture | in 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Department of Neurosurgery Charité Berlin, Berlin, Germany
- Buda Health Center, Budapest, Hungary
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No